CLINICAL TRIAL: NCT05619159
Title: the Value of Immunohistochemical Expression of Moesin in Endometrial Hyperplasia and Endometrial Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nermin Abbas, resident doctor pathology in sohag oncology center, Sohag University
Other Study IDs: Soh-Med-22-10-04
Record Dates: First submitted 2022-10-23; First posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Endometrial Cancer and Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Neoplasms; Endometrial Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endometrial carcinoma smples
  Interventions: Device: microscopic pathological evaluation
- endometrial hyperplasia samples
  Interventions: Device: microscopic pathological evaluation

INTERVENTIONS:
Device: microscopic pathological evaluation — description of moesin expression between endometrial hyperplasia and endometrial carcinoma

SUMMARY:
Endometrial carcinoma (EC) is the most prevalent invasive carcinoma of the female genital tract in developed countries, while it ranks as the second most frequently occurring neoplasm of women in developing countries, after carcinoma of the cervix uteri. The vast majority of ECs occur in perimenopausal and postmenopausal women .

ECs are classified into two distinct phenotypes; type I which represents more than 80% of all cases of ECs, it has a favorable prognosis. This type is linked to excess, unopposed hyper-estrogenic condition and it is almost always preceded by endometrial hyperplasia. On the contrary, type II endometrial carcinoma is less common than type I, representing less than 10% of all cases of ECs. Type II endometrial carcinomas are high grade, poorly differentiated and estrogen-independent tumors .

ELIGIBILITY:
Inclusion Criteria:

* Hysterectomy specimens diagnosed as endometrial hyperplasia and endometrial adenocarcinoma.
* All cases of endometrial biopsies obtained by curettage (D&C) diagnosed as endometrial hyperplasia.
* Cases of cyclical endometrium obtained from endometrial curettage or hysterectomy specimens done for pathological conditions other than hyperplastic or neoplastic endometrial lesions.
* Complete clinical data.

Exclusion Criteria:

* Patients with a history of preoperative chemotherapy and /or radiotherapy.
* Biopsies with predominantly blood clots.
* Insufficient or tiny tissue biopsies.

Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: females presented to gynecology department in sohag university hospital and sohag oncology center
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
The value of immunohistochemical expression of moesin in endometrial hyperplasia and endometrial carcinoma | 1 year
  To evaluate immunohistochemical expression of moesin in normal, hyperplasic and neoplastic endometrial tissues , correlate this expression with different clinicopathologic parameters of endometrial carcinoma and to evaluate the role of moesin as prognostic marker in progression from preinvasive lesions of the endometrium to endometrial carcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frose J, Chen MB, Hebron KE, Reinhardt F, Hajal C, Zijlstra A, Kamm RD, Weinberg RA. Epithelial-Mesenchymal Transition Induces Podocalyxin to Promote Extravasation via Ezrin Signaling. Cell Rep. 2018 Jul 24;24(4):962-972. doi: 10.1016/j.celrep.2018.06.092. PMID 30044991
- [Background] Wang H, Xiao X, Li Z, Luo S, Hu L, Yi H, Xiang R, Zhu Y, Wang Y, Zhu L, Xiao L, Dai C, Aziz A, Yuan L, Cui Y, Li R, Gong F, Liu X, Liang L, Peng H, Zhou H, Liu J. Polyphyllin VII, a novel moesin inhibitor, suppresses cell growth and overcomes bortezomib resistance in multiple myeloma. Cancer Lett. 2022 Jul 1;537:215647. doi: 10.1016/j.canlet.2022.215647. Epub 2022 Mar 17. PMID 35306105
- [Background] Mandelbaum RS, Ciccone MA, Nusbaum DJ, Khoshchehreh M, Purswani H, Morocco EB, Smith MB, Matsuzaki S, Dancz CE, Ozel B, Roman LD, Paulson RJ, Matsuo K. Progestin therapy for obese women with complex atypical hyperplasia: levonorgestrel-releasing intrauterine device vs systemic therapy. Am J Obstet Gynecol. 2020 Jul;223(1):103.e1-103.e13. doi: 10.1016/j.ajog.2019.12.273. Epub 2020 Jan 21. PMID 31978437
- [Background] Yuan O, Ugale A, de Marchi T, Anthonydhason V, Konturek-Ciesla A, Wan H, Eldeeb M, Drabe C, Jassinskaja M, Hansson J, Hidalgo I, Velasco-Hernandez T, Cammenga J, Magee JA, Nimeus E, Bryder D. A somatic mutation in moesin drives progression into acute myeloid leukemia. Sci Adv. 2022 Apr 22;8(16):eabm9987. doi: 10.1126/sciadv.abm9987. Epub 2022 Apr 20. PMID 35442741